CLINICAL TRIAL: NCT05508113
Title: Effects of Ozone Autohemotherapy on Patients With Post-ischemic Stroke Insomnia
Brief Title: Ozone Autohemotherapy for Ischemic Stroke Sleep Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mengmeng Chen (Other)
Responsible Party: Sponsor-Investigator, Mengmeng Chen, Principal Investigator, Jilin University
Organization: Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2022100
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Post-ischemic Stroke Insomnia
Keywords: Ischemic stroke; Insomnia; Ozone Autohemotherapy
MeSH Terms: conditions — Ischemic Stroke; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention was given to this group of patients
- 20-40ug/ml ozone (Experimental): ozone autohemotherapy
  Interventions: Other: ozone autohemotherapy

INTERVENTIONS:
Other: ozone autohemotherapy — After autologous blood is mixed with ozone in vitro, the blood is injected into the patient through intravenous infusion
  Arms: 20-40ug/ml ozone

SUMMARY:
The purpose of this study is to observe the efficacy and safety of ozonated autohemotherapy in patients of post-ischemic stroke insomnia and to explore its mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria for ischemic stroke; Insomnia quality index (ISI) score > 7 points

Exclusion Criteria:

* acute ischemic stroke; associated with failure of important organs or malignant tumor; patients with worsening condition, new cerebral infarction or secondary cerebral hemorrhage; with comprehension or cognitive impairment, unable to fully understand the scale and unable to cooperate with treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-26 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | 2 weeks
  The Insomnia Severity Index Scale (ISI) will be used, which scale ranges from 0 to 28, with higher scores representing more severe insomnia. Specifically, 0-5 points represent excellent sleep quality, 6-10 points mean good sleep quality, 11-15 points indicate average sleep quality, and 16-21 points represent poor sleep quality.
Pittsburgh Sleep Quality Index | 2 weeks
  The Pittsburgh Sleep Quality Index Scale (PSQI) will be used, which scale ranges from 0 to 21, with higher scores representing poorer sleep quality. In detail, 0-7 points represent insomnia of no clinical significance, 8-14 points mean sub-clinical insomnia, 15-21 points indicate moderate clinical insomnia, and 22-28 points represent severe clinical insomnia.

SECONDARY OUTCOMES:
brain-derived neurotrophic factor (BDNF) | 2 weeks
  Detection of BDNF in serum of patients using Elisa kit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sekerdag E, Solaroglu I, Gursoy-Ozdemir Y. Cell Death Mechanisms in Stroke and Novel Molecular and Cellular Treatment Options. Curr Neuropharmacol. 2018;16(9):1396-1415. doi: 10.2174/1570159X16666180302115544. PMID 29512465
- [Background] Masan J, Sramka M, Rabarova D. The possibilities of using the effects of ozone therapy in neurology. Neuro Endocrinol Lett. 2021 Mar;42(1):13-21. PMID 33932964
- [Background] Kadir K, Syam Y, Yusuf S, Zainuddin M. Ozone Therapy on Reduction of Bacterial Colonies and Acceleration of Diabetic Foot Ulcer Healing. Home Healthc Now. 2020 Jul/Aug;38(4):215-220. doi: 10.1097/NHH.0000000000000889. PMID 32618780
- [Background] Martinez-Sanchez G, Delgado-Roche L, Diaz-Batista A, Perez-Davison G, Re L. Effects of ozone therapy on haemostatic and oxidative stress index in coronary artery disease. Eur J Pharmacol. 2012 Sep 15;691(1-3):156-62. doi: 10.1016/j.ejphar.2012.07.010. Epub 2012 Jul 13. PMID 22796450